CLINICAL TRIAL: NCT00417287
Title: A Randomized Phase II Open-Label Study of Two Different Dose Levels of PX-12 in Patients With Advanced Carcinoma of the Pancreas Whose Tumors Have Progressed on Gemcitabine or on a Gemcitabine-Containing Combination
Brief Title: Phase II Study of PX-12 in Patients With Advanced Pancreatic Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Investigator decision
Sponsor: Cascadian Therapeutics Inc. (Industry)
Collaborators: National Cancer Institute (NCI) (NIH); Translational Genomics Research Institute (Other)
Responsible Party: Sponsor
Organization: Seagen Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PX-12-II-01; P01CA109552 (NIH)
Record Dates: First submitted 2006-12-29; First posted 2007-01-01 (Estimated); Last update posted 2018-05-16 (Actual); Status verified 2015-04

CONDITIONS: Pancreatic Neoplasms
Keywords: Pancreas; Cancer; Carcinoma
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasms; Carcinoma | interventions — thioredoxin reductase inhibitor AM12

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High dose (Active Comparator): 128 mg/m2
  Interventions: Drug: PX-12
- Low dose (Active Comparator): 54 mg/m2
  Interventions: Drug: PX-12

INTERVENTIONS:
Drug: PX-12 — 3 hour intravenous infusion as a dose of either 54 mg/m2 or 128 mg/m2 daily for 5 days every three weeks.
  Other Names: Thioredoxin Inhibitor

SUMMARY:
This study is being conducted to evaluate the clinical efficacy, biologic activity (inhibition of PX-12 target thioredoxin-1) and effects of an expired metabolite of PX-12 in patients with advanced pancreatic cancer.

DETAILED DESCRIPTION:
In a Phase I trial, PX-12 demonstrated anti-tumor activity and pharmacodynamic activity across a wide dose range. At higher doses, one side effect of the agent was a garlic-like odor of an expired metabolite. This study is being conducted to evaluate the clinical efficacy, biologic activity (inhibition of PX-12 target thioredoxin-1) and effects of the expired metabolite at two dose levels of PX-12. This study will determine if the efficacy and biologic activity achieved at either of the two dose levels is sufficient to proceed to further studies without pushing to the maximally tolerated dose.

ELIGIBILITY:
Inclusion Criteria:

* Histologically- or cytologically-confirmed diagnosis of advanced carcinoma of the pancreas (stage IV disease only).
* Patients whose tumor has progressed on gemcitabine or on a gemcitabine-containing combination. Patients must have received no more than two prior regimens for metastatic disease. Use of gemcitabine as a radiation sensitizer in combination with radiotherapy for localized disease will not be considered a prior gemcitabine-containing regimen if gemcitabine was received for ≤ 1 month following completion of radiotherapy. In addition, the use of 5-fluorouracil as a radiation sensitizer for localized disease will be allowed and not counted as a prior regimen if the 5-FU was continued for ≤ 1month following completion of radiotherapy.
* Karnofsky Performance Status of ≥ 70%.
* Patients must have discontinued previous anti-cancer therapy or other investigational agent at least three weeks or within 5 half lives of the drug (whichever is shorter) prior to entry into the study (six weeks for mitomycin C or nitrosureas) provided that all toxicities from prior treatment have resolved to a Grade 1 or less.
* Patients must have discontinued radiation therapy at least two weeks prior to entry into the study and have recovered from all radiation-related toxicities.
* Adequate organ function including the following:
* ANC ≥ 1500 cells/microL; platelets > 100,000/microL; hemoglobin ≥ 9 g/dL (may be transfused to this level).
* Bilirubin ≤ 2.0 mg/dL; aspartate transaminase (AST/SGOT) and alanine transaminase (ALT/SGPT) ≤ 3.0 times institutional upper limit of normal (ULN) OR < 5 times institutional ULN if the subject has documented liver metastases.
* Creatinine ≤2.0 mg/dL.
* CA19-9 level >2 times ULN.
* Disease that is measurable by CT scan per RECIST criteria (Appendix IV).
* PET/CT or PET scan with SUV of ≥ 5.0 in at least one lesion on an 18F FDG scan.

Exclusion Criteria:

* Active infection requiring antibiotics at study entry.
* Any serious concomitant systemic disorder that in the opinion of the investigator would place the patient at excessive or unacceptable risk of toxicity.
* Patients with active (requiring continuous medical therapy) pulmonary disease (COPD, asthma) or evidence of interstitial pneumonitis or pulmonary fibrosis on baseline chest X-ray or PET/CT scan.
* Significant central nervous system or psychiatric disorder(s) that preclude the ability of the patient to provide informed consent.
* Known or suspected brain metastases that have not received adequate therapy. Patients must be stable without requirement for steroids or seizure medications.
* Major surgery within 4 weeks of study entry.
* Chemotherapy/investigational drugs within 3 weeks or within 5 half lives of the drug (whichever is shorter) of study entry, provided that all toxicities from prior treatment have resolved to a Grade 1 or less.
* Inability to tolerate prophylactic (1 mg/day) coumadin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2006-12; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Progression free survival and overall survival (percentage of patients alive at 6 months) | 6 months
Determine if there is a difference in effect on circulating Trx-1 protein levels between two dose levels of PX-12 | 21 days

SECONDARY OUTCOMES:
Determine which of two dose levels of PX-12 causes the greatest effect on three surrogate markers of clinical activity | 42 days
Determine effects of two different dose levels on overall clinical response | 42 days
Further evaluate safety profile of PX-12 | 21 days
Assess the effects of metabolic excretion of PX-12 | 3 hours

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - TGen Clinical Research Services at Scottsdale Healthcare, Scottsdale, Arizona
  - Arizona Cancer Center, University of Arizona, Tucson, Arizona
  - The University of Texas M.D. Anderson Cancer Center, Houston, Texas